CLINICAL TRIAL: NCT03898128
Title: ItaliaN Observational Study of Patients With Acute Lymphoblastic Leukemia Treated With Anti-CD22 Immunoconjugate
Acronym: INO-CD22
Status: Completed | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRST204.03
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anti-CD22 Immunotoxin — Clinical data (treatment, survival, adverse events) of patients treated with anti-CD22 immunoconjugates from 2014 will be collected

SUMMARY:
In phase 2 and phase 3 studies, inotuzumab has shown evidence of single agent anti-leukemic activity and proved to be particularly effective in providing a deep response, with an acceptable safety profile. Since 2014 anti-CD22 has been available for compassionate use in Italy.

In this non-interventional retrospective study, toxicity, effectiveness and costs assessment data will be collected from patients with ALL, to improve the knowledge about anti-CD22 treatment in clinical practice. Collecting data of patients and analyzing a large unbiased patient-set of patients receiving anti-CD22 immunoconjugates could enlarge our knowledge on therapies engaging CD22

DETAILED DESCRIPTION:
In phase 2 and phase 3 studies, inotuzumab has shown evidence of single agent anti-leukemic activity and proved to be particularly effective in providing a deep response, with an acceptable safety profile. Since 2014 anti-CD22 has been available for compassionate use in Italy.

In this non-interventional retrospective study, toxicity, effectiveness and costs assessment data will be collected from patients with ALL, to improve the knowledge about anti-CD22 treatment in clinical practice.

Despite recent advancements in the treatment of hematological malignancies, still a considerable number of cases cannot be cured and represent real societal challenges with a relevant social and economic impact. Indeed, treatments are becoming more expensive and the current state of the art does not allow a good prediction of the therapeutic outcome. In particular, several steps of the diagnostic and therapeutic paths should be improved, from early and advanced diagnosis, in order to avoid treatment delays or impairment, to prognostic assessment and monitoring of therapeutic response. The unsatisfactory response to conventional chemotherapy has led to the development of high-cost targeted therapies, whose administration and schedules has to be guided by defined molecular criteria. Beside the economic perspective, these novel drugs have relevant side effects that cannot be predicted before treatment starts.

The management of hematological malignancies is further complicated by the high level of disease heterogeneity in terms of pathogenetic and molecular mechanisms. A number of subtypes have been defined for each disease, based on cytogenetic and molecular profiles and relevant differences can be even observed within the same disease subtype, leading to different clinical outcomes and responses to treatment and to guide therapeutic decisions for patients affected by CD22 positive ALL.

Due to the observational nature of the study, for the patient there is no benefit expected. For this observational nature of the study, for the patient there is no risk about his health. Data will be treated according GCP/EU laws/Italian laws/local laws according the most restrictive between these laws.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with ALL according WHO 2016 classification.
2. Patient who received any anti-CD22 immunoconjugate from 2014 to 01-Mar-2019 outside clinical trials.

Exclusion Criteria:

1. Patients who received anti-CD22 treatment within a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALL patients treated with anti-CD22 immunoconjugate drugs from 1-Jan-2014 to 01-Mar-2019
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events of grade 3 and 4 | up to 12 months
  toxicity profile of the therapy with antiCD22 immunoconjugates in patients with ALL

SECONDARY OUTCOMES:
Overall survival | up to 18 months
  Overall Survival (OS), defined as the number of days between the first study drug administration and death from any cause
Disease free survival | up to 18 months
  Disease Free Survival (DFS), defined as the number of days between the first study drug administration and any event including disease progression or death from any cause
Response to therapy | up to 18 months
  response to therapy (CR, CRi, MRD and bridge to transplant)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, Prof, Study Director — IRST IRCCS; Delia Cangini, MD, Principal Investigator — IRST IRCCS
Locations (5):
- Italy (5):
  - Irst Irccs, Meldola (FC), FC
  - AUSL Romagna, Ravenna, RA
  - Azienda ULSS2 Marca Trevigiana, Treviso, TV
  - ULSS 3 Serenissima, Mestre, Venezia
  - Ospedale S. Eugenio, Roma